CLINICAL TRIAL: NCT05270148
Title: High-intensity Interval Training Versus Fatmax Training in Diabetic Type 2
Acronym: Lipidox
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Cadiz (Other)
Collaborators: Instituto de investigación e innovación biomédica de Cádiz (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Lipidox
Record Dates: First submitted 2021-12-17; First posted 2022-03-08 (Actual); Last update posted 2022-11-03 (Actual); Status verified 2022-10

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: HIIT; Fatmax; Maximum Fat oxidation; Diabetes Mellitus 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Intervention Model Description: Randomized Control Trial
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- HIIT Group (Experimental): Participants are enrolled in a high-intensity interval training exercise program
  Interventions: Other: HIIT
- FatMax Group (Active Comparator): Participants who are enrolled in a moderate-intensity continuous training exercise program
  Interventions: Other: Fat Max
- Control (No Intervention): Participants who do not receive an exercise program. They will be instructed to maintain their normal life habits with respect to physical activity and diet.

INTERVENTIONS:
Other: HIIT — 12 weeks training High-Intensity Interval Training consists of 3 sessions per week in a cycle ergometer, with 1-2days off between sessions, under the supervision of a personal trainer. HIIT program will consist of 3-5 series of 1 min duration at 90-130% of its maximum power (determined in the first training session), with 90 seconds of rest between sets (estimated total time of the session: 10 minutes).Depending on the number of training session, the loadand the series will increase up to 40% more than the maximum load.
  Arms: HIIT Group
Other: Fat Max — 12 weeks training Fatmax consist in 3 sessions per week in a cycle ergometer, with 1-2days off between sessions, under the supervision of a personal trainer. MICTprogram will consist of sessions of approximately ˜45min of moderate aerobic exercise (at the intensity at which the maximal fat oxidation was achieved in the laboratory test) in cycle ergometer.
  Arms: FatMax Group

SUMMARY:
The project investigates the effects of two exercise protocols at different intensities, high-intensity interval training and constant load at Fatmax, for 12 weeks in maximal fat oxidation, hormonal regulation of appetite, and insulin sensitivity in persons with obesity and type 2 diabetes mellitus. The participants will be of both sexes with ages between 40 and 55 years, belonging to the Province of Cádiz. Sixty volunteers will be randomly allocated into three groups: High-Intensity Interval TRaining (HIIT), Fatmax, and control groups. The assessments will be at the previous exercise intervention, posterior the exercise intervention, and 12 weeks after the last intervention. The outcome variables will include body composition, oral glucose tolerance test, appetite, plasma glucose, lipids in plasma, hormones, and adipokines.

ELIGIBILITY:
Inclusion Criteria:

* Non-smoking
* Non-alcoholic (<3 standard drinks per day)•Body mass index >25 kg/m maintaining the habitual dietary patterns without a body mass reduction higher than 2% during the last 6 months
* Not being insulin dependent
* Absence of injury, disease or disability or other known medical condition which could affect the ability to successfully participate in physical exercise tests
* Absence of cardiovascular disease (angina, peripheral or cerebro-vascular disease, etc.).
* Absence of neurologic and psychiatric diseases.
* Absence of respiratory diseases (pulmonary hypertension, chronic obstructive pulmonary disease, etc.).
* Absence of other metabolic diseases (hyper/hypoparathyroidism, hyper/hypothyroidism, Cushing's disease, Type 1 diabetes, etc.)
* Absence of active inflammatory bowel disease
* Absence of kidney disease
* Absence of tumors
* Absence of coagulation dysfunction
* Not under treatment with medications k known to affect glucose metabolism, recent steroid treatment (within 6 months), or hormone replacement therapy
* Be able to understand communication in Spanish or English.

Exclusion Criteria:

* They do not attend more than 2 or 4 consecutive sessions of nutritional counseling or physical training respectively.
* Missing more than 4 or 6 sessions in total of nutritional counseling or physical training respectively.

Ages: 40 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-03-10 (Actual); Primary Completion 2023-09-01 (Estimated); Study Completion 2024-08-31 (Estimated)

PRIMARY OUTCOMES:
Maximal fat oxidation (MFO) | 12 weeks
  Maximal fat oxidation test (MFO) to determine the maximal fat oxidation during exercise (MFO), a gradual test on cycloergometer (Lode Excalibur, Netherlands) will be performed. The test will begin with a load of 15 Watts, increasing 15Watts every 3 minutes until the respiratory quotient reaches a stable value of 1 or higher. Throughout the test a cadence of 80 r.p.m. will be maintained. Calculation in the base of expired gases will be made for the estimation of grams per minute of fat oxidation.
Cardiorespiratory fitness | 12 weeks
  The maximal oxygen consumption (VO2max) during exercise in liters per minute by a gradual test on a cycle ergometer (Lode Excalibur, Netherlands) will be performed. The gas exchange will be measured by Jaeger MasterScreen CPX® (CareFusion, San Diego, USA)The test will be continuing the MFO from the load when the respiratory quotient reaches a stable value of 1 or higher. Once this point is reached, 15 Watts increments will occur every minute until exhaustion is reached, until achieving the VO2max. Throughout the test a cadence of 80 r.p.m. will be maintained. Heart rate will be recorded in beats per minute.
Blood samples | 12 weeks
  Glucose and insulin concentrations will be determined using ELISA technique and will be combined to report the Homeostatic Model Assessment for Insulin Resistance (HOMA-IR) insulin sensitivity index will be calculated
Appetite assessment | 12 weeks
  Since appetite feeling modulate nutritional behaviour, the evaluation of appetite among the intervention groups can improve the quality of the study from a comprehensive perspective. After a period of 8-10 hours of fasting, an analog visual scale (AVS) will be completed in order to ensure the appetite felt by the participant in the morning. The AVS runs from 1 to 10, being the lowest value no appetite at all, and the maximum full appetite.
Body composition: Fatmass and Fat-free mass. | 12 weeks
  Body composition will be estimated using a multifrequency bioimpedance of 8 electrodes previously validated (TANITAMC780MA). The calculation of impedance can estimate the fat mass and fat-free mass in kilograms. The patients will wear light clothing and will assume a posture in accordance with the manufacturers' instructions. Other previous considerations will be followed 24 hours before the measure: (i) to refrain from vigorous exercise, (ii) to take alcoholic drinks, (iii) to take energy drinks, and (iv) to be in a fasting state for at least 8 hours. Hydration status will be controlled through a urine color scale from clear to dark during the 7 days before assessment for adjusting variables.

SECONDARY OUTCOMES:
Accelerometry | 12 weeks
  Physical activity assessment will be carried out through accelerometers (direct method) at the wrist during 7consecutive days. The data generated by the accelerometers will be analysed by using ActiLife 6.6.2 software (ActiGraph, Florida; USA), using Freedson (1998) cut-points for adults and Choi's validation. The software calculates in the base the movements of the accelerometer's time of light, moderate, and vigorous physical activity in minutes.
Assessed changes from physical activity | 12 weeks
  Physical activity assessment will be estimated by the participant's self-reported International Physical Activity Questionnaire Short Version (IPAQ-SF) previously validated in Spain. The IPAQ-SF estimates the sedentary time, moderate and vigorous activity time in minutes per week. The questionnaire made a classification in high physical activity level (>3000 of the metabolic equivalent of task (MET) minute per week in moderate or >1500 MET min/week in vigorous activity), moderate physical activity level (>600 MET min/week of moderate or vigorous activity), and low activity level (<600 MET min/week of moderate or vigorous activity)
Blood pressure | 12 weeks
  Systolic and diastolic blood pressures will be recorded three times by using the validated bloodpressure monitoring device with the participant seated, back supported in chair and feet flat on floor without legscrossed, after they rested 5 minutes. The guidelines of the Hypertension and Cardiology European Societies and the Spanish one will be used to classify blood pressure stages of participants.
Self-reported quality of life | 12 weeks
  Self-reported quality of life will be registered by applying the Short Form 36-health survey (SF-36) questionnaire previously validated in Spain. The SF-36 is a generic measure of quality of life and has been evaluated for a wide variety of medical conditions, including diabetes. The SF-36 includes 36 questions that evaluate 8 subscales, scores for each scale range from 0 to 100, with higher scores indicating a higher level of function or wellbeing. The physical component summary is derived from the 4 subscales of physical functioning, role physical, bodily pain, and general health; while the mental component summary is derived from the subscales of vitality, social functioning, role emotional, and mental health.

CONTACTS AND LOCATIONS:
Overall Officials: Jesús Ponce, PhD, Principal Investigator — University of Cadiz
Locations (1):
- Science of Education Faculty, Puerto Real, Cadiz, Spain

IPD SHARING:
Plan to Share IPD: No